CLINICAL TRIAL: NCT05646680
Title: A Performance Study of (Opportunistic) Salpingectomy
Acronym: QOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-11611
Record Dates: First submitted 2022-11-24; First posted 2022-12-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Adnexal Lesion; Ovarian Cancer
Keywords: salpingectomy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- two step adnexectomy (Other): Patients planned for unilateral or bilateral adnexectomy (removal of ovary and salpinx) will have their adnexectomy performed in two steps in the same surgical episode: first the salpingectomy (removal of the salpinx), then the oophorectomy (the removal of the ovary).
  Interventions: Procedure: two step adnexectomy

INTERVENTIONS:
Procedure: two step adnexectomy — instead of standard resection of salpinx and ovary, they are now separately excised

SUMMARY:
The goal of this clinical trial is to test the quality of the performance of opportunistic salpingectomies in women scheduled for adnexectomy. The main questions it aims to answer are:

* How many salpingectomies are incomplete?
* Are there any factors related to incomplete resection? Could the investigators develop a instruction video to optimize the surgical technique?

Participants planned for uni-or bilateral adnexectomy (removal of ovary and salpinx) will have their adnexectomy in two steps in the same surgical episode: first the salpingectomy (removal of the salpinx), then the oophorectomy (the removal of the ovary).

DETAILED DESCRIPTION:
Rationale: Salpingectomy in post-reproductive women could reduce the risk of developing ovarian cancer. In women at high risk for ovarian cancer (because of genetic mutations) a risk reducing salpingectomy with delayed ovariectomy could be an advantage. It is considered that salpingectomy does not cause premature menopausal symptoms. Prospective randomized trials are being performed to estimate the true risk reducing effect of salpingectomy on ovarian cancer. Those studies are based on a complete bilateral salpingectomy.

Objective: The QOS study investigates the quality of performance of opportunistic salpingectomy and the risk factors associated with reminiscing fimbrial tissue after salpingectomy.

Study design: Multicenter interventional trial

Study population: Patients planned for unilateral or bilateral adnexectomy (removal of ovary and salpinx) will be counselled to participate.

Intervention: The gynecologist will perform the adnexectomy in two steps in the same surgical episode: first the salpingectomy (removal of the salpinx), then the oophorectomy (the removal of the ovary). The pathologist investigates for pathology and describes if fimbrial tissue (the last part of the salpinx adjacent to the ovary) has been left behind on the ovarian surface microscopically and macroscopically.

Main study parameters/endpoints: The primary outcome is the percentage of incomplete salpingectomies. Secondary outcome is the detection of factors related to incomplete resection of the salpinx. If necessary a guideline/instruction video could be developed to optimize the surgical technique. A total of 200 specimens are to be included to answer the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for uni- or bilateral adnexectomy. (may be in combination with hysterectomy) AND * competent to act on itself

* dutch speaking
* signed informed consent

Exclusion Criteria:

* Endometrial cancer or invasive cervical cancer

* radiotherapy in the pelvis in the medical history
* (partial) salpingectomy
* Pelvic Inflammatory Disease
* Adnexectomy for gender transformation surgery if wish to preserve the ovarian tissue.
* Surgery in two steps is not safe to perform
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only female patients receive hysterectomy
Enrollment: 115 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Percentage of incomplete salpingectomies | 10 days
  The rate of ovarian samples on which residual fimbrial or fallopian tube tissue has been left behind.(macroscopically and microscopically)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Ghent, Belgium